CLINICAL TRIAL: NCT04664608
Title: Evaluation of a Wireless EEG Monitor for Pediatric Patients
Brief Title: Pediatric EEG Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: 2020-3266
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pediatric ALL; Epilepsy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: wearable EEG sensor — Wireless wearable EEG devices offer a new, non-invasive, and easy way of performing EEG monitoring.

SUMMARY:
The purpose of this study is to understand if a new, smart, wireless EEG developed by our team can be used to monitor the continuous electrical activity of the brain in the ICU and EMU and whether it works as well as the current standard, wired EEGs.

DETAILED DESCRIPTION:
The investigators propose to 1) optimize these devices for use in pediatric ICU patients, 2) demonstrate safety, reliability, and accuracy of these devices for continuous ICU EEG signal measurements, and 3) demonstrate these devices are preferred by patients and parents to current EEG devices. Once validated, such sensors could fundamentally change the way patients are monitored by EEG in the ICU, allowing wireless, continuous, real-time detection of brain wave activity in ICU patients, reducing limitations in mobility as well as access by staff and caregivers to the patient, and ultimately offering opportunity to reduce morbidity and mortality in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be admitted to the PICU or EMU at Lurie Children's and are prescribed an EEG as part of their standard of care.

Exclusion Criteria:

* Anyone with a skin abnormality that would potentially increase the risk of device use will be excluded.
* Ages 18 years or older.
* Any patient or family determined by an attending physician or bedside care team to be too unstable (patient) or experiencing too much stress (family) will not be approached for recruitment.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children between the ages of 0 and 18 years of age who are prescribed an EEG while admitted to the pediatric intensive care unit (PICU) or Epilepsy Monitoring Unit (EMU)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Percent Agreement | 3 years
  Percent agreement between experimental sensor and commercially available electroencephalogram (EEG)

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States